CLINICAL TRIAL: NCT04131465
Title: Home HIV Testing for Older Adults and Their Family and Community Members: a Three-arm Randomized Controlled Trial in Rural South Africa
Brief Title: Home HIV Testing for Older Adults in South Africa
Acronym: Test@Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: University of Heidelberg Medical Center (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Till Barnighausen, Adjunct Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NIH/NIA- 2P01AG041710-04
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections; Knowledge, Attitudes, Practice
Keywords: HIV testing; HIV status knowledge; Health system; Community health workers
MeSH Terms: conditions — HIV Infections; Behavior

STUDY DESIGN:
Intervention Model Description: This study will randomize older adults living in a rural community in South Africa to one of three trial arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessors will not know the arm assignment when they assess the outcomes. The investigators analyzing the data for the initial effect size estimations will be blinded to the arm assignment. Care providers (i.e., the fieldworkers providing the home-based HIV testing) and participants cannot be blinded to the assignment to the trial arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home HIV self-testing (Experimental): Fieldworkers will visit potential participants in their homes and offer 3 oral HIV self-testing kits with a short introduction to HIV self-testing.
  Interventions: Diagnostic Test: Home HIV self-testing
- Home HIV rapid testing (Experimental): Fieldworkers will visit potential participants in their homes and offer home-based HIV rapid testing and counselling.
  Interventions: Diagnostic Test: Home HIV rapid testing
- Home HIV self-testing and rapid testing (Experimental): Fieldworkers will visit participants in their homes and offer 3 oral HIV self-testing kits with a short introduction to HIV self-testing as well as home-based HIV rapid testing and counselling.
  Interventions: Diagnostic Test: Home HIV self-testing and rapid testing

INTERVENTIONS:
Diagnostic Test: Home HIV self-testing — Offer of 3 OraQuick HIV self-test kits
  Arms: Home HIV self-testing
Diagnostic Test: Home HIV rapid testing — Offer of HIV rapid testing with Alere Determine HIV-1/2
  Arms: Home HIV rapid testing
Diagnostic Test: Home HIV self-testing and rapid testing — Offer of 3 OraQuick HIV self-test kits and HIV rapid testing with Alere Determine HIV-1/2
  Arms: Home HIV self-testing and rapid testing

SUMMARY:
Many older adults in rural South Africa still lack knowledge of their HIV status despite a high probability of infection. Older adults tend to test less for HIV because most HIV testing and prevention programs have been targeted at younger age groups. Other reasons for failure to test for HIV include frailty and lack of financial resources to travel to HIV testing centers. Home-based testing is a powerful approach to bring HIV testing services -- and HIV status knowledge -- to older adults. In real-life health systems, community health workers, such as the South African community care givers, could potentially provide home-based HIV testing on a routine basis. In this study, the investigators are trying to establish the best 'form' for the 'function' home-based HIV testing.

Specifically, the investigators aim to

1. Establish the comparative effectiveness of three home-based HIV testing options among older adults in rural South Africa
2. Identify spill-over effects of the different home-based HIV testing options to other adults in the households and communities of the older adults receiving the testing options
3. Determine the comparative cost-effectiveness of the three home-based HIV testing options among older adults.

DETAILED DESCRIPTION:
Background In the first wave of a large population-representative study of older adults in rural South Africa, the 'Health and Aging in Africa: A Longitudinal Study of an INDEPTH Community in South Africa (HAALSI)' study, large gaps in knowledge of HIV status were found among participants, coupled with low rates of recent HIV testing and high rates of sexual behaviour that can lead to acquisition and transmission of HIV. In general, older adults should test for HIV at least once per year (HIVAge.org), but few do so, in part because current HIV testing programmes have traditionally focused on young and middle-age adults and HIV testing facilities are often difficult to access for older populations. Only 17% of older adults in the HAALSI community reported having tested for HIV in the past 6 months.

Home testing can provide a powerful approach to bring the health systems 'function' of HIV testing to older adults in rural Africa. In the routine health system, community health workers, such as the South African community care givers, could provide this 'function' on a regular basis. Home rapid HIV testing and HIV self-test kits have been intensively studied in many populations. HIV self-test kits have recently become available as over the- counter products in South Africa, after the South African Pharmacy Council (SAPC) lifted a ban on their sale in pharmacies in December 2016.

To date, however, no study has compared head-to-head different 'forms' of home testing for HIV. In this study, the investigators aim to establish the comparative effectiveness and cost-effectiveness of three different options of home HIV testing among older adults in rural South Africa: (1) home delivery of HIV self-test kits, (2) home HIV rapid testing, and (3) both home delivery of HIV self-test kits and home HIV rapid testing.

Overall, home HIV testing is likely attractive for older adults because it allows testing without having to visit a health care facility. Home delivery of HIV self-testing kits has the additional advantage that it allows HIV testing in a place and at a time of one's own choosing. Home approaches to HIV testing are particularly policy-relevant at this time, because South Africa and many other countries in sub-Saharan Africa are currently expanding in re-designing their community health worker programs, through which home HIV testing could be provided on a routine basis.

Preliminary evidence in this and in other populations have suggested that HIV testing and linkage to HIV treatment and care improve health care utilization for other non-HIV chronic care and reduce risky sexual behavior. The investigators will thus not only assess the effects of the different home HIV testing offers on HIV testing but also assess comparative effects on healthcare utilization, noncommunicable disease endpoints, and sexual behaviors.

Research Aims

This study thus aims to:

1. Establish the comparative effectiveness of three options for home HIV testing for older adults in rural South Africa
2. Identify spill-over effects of the different options for home HIV testing to other adults in the families and communities of the older adults receiving the testing options
3. Establish the comparative cost-effectiveness of the three options for home HIV testing among older adults.

Study Design Participants in Wave 2 of the HAALSI study will be offered one of three options (randomly assigned 1:1:1) for home HIV testing: (1) three oral HIV self-test kits with a brief introduction to HIV self-testing (home HIV self-testing arm), (2) home rapid HIV testing and counselling (home rapid HIV testing arm), and (3) three oral HIV self-test kits with a brief introduction to HIV self-testing plus home rapid HIV testing and counselling (home HIV self-testing and HIV rapid testing arm). The brief introduction to HIV self-testing will include encouragement of both self-use and onward distribution to household and community members.

The HAALSI participants were randomized (sample ~3,600; 1,200 individuals in each of the three arms). Randomization has occurred during routine HAALSI fieldwork visits, using a pre-programmed randomization process that is integrated into the tablet-based HAALSI computer-assisted personal interview (CAPI). This randomization was completed during a three-month period between May and July 2019.

Outcome Assessment The primary outcomes (1-2) and a group of secondary outcomes (3-21) will be assessed by telephone at 9 months after randomization. Based on the timing of randomization, primary data collection will take place from February through May 2020. Then, both the primary and an expanded set of secondary outcomes including several biologically-measured secondary outcomes (1-25) will be assessed at 18-24 months, during the subsequent, planned cohort-based data collection (HAALSI Wave 3).

Power Calculation In the first wave of the HAALSI study, the proportion of people having tested for HIV in the past 6 months (which was about 17%) was measured. Assuming uniform distribution of testing over time, it would be expected that about 3% of older adults in the HAALSI population tested in the past month. Based on the HAALSI 1 data, the proportion of older adults who ever tested for HIV is 65%. Given these estimates for the endpoints in the control arm, this study is powered to detect a 3 percentage point difference in HIV testing in the past month and a 6 percentage point difference in ever testing for HIV across the three arms. For this power calculation the investigators further assumed, 20% loss to follow-up, 80% power and a significance level for rejecting the Null hypothesis of 0.0167. This significance level results from the adjustment of the standard 0.05 significance level for multiple hypothesis testing - each arm compared to each other arm - using the Holm-Bonferroni method.

Data Analyses The investigators will measure risk ratios for all the binary outcomes in this study, using modified Poisson regression implemented in generalized linear models with Poisson distribution and log link. Furthermore, the effect sizes for count outcomes using generalized linear models with negative binomial distribution and log link will be measured; the investigators will measure effect sizes for continuous outcomes using generalized linear models with normal distribution and identity link. All estimations will be adjusted for clustering of outcomes at the household level as well as for baseline values of the endpoints. Baseline values of our primary and secondary endpoints will be assessed during the baseline visit before the HAALSI participants receive the trial exposure.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be part of the second wave of a population-representative longitudinal study in rural South Africa: "Health and Aging in Africa: A Longitudinal Study of an INDEPTH community in South Africa" (HAALSI)
* Mental capacity to consent to participation in this study

Exclusion Criteria:

* Participants who meet the inclusion criteria but do not wish to participate in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3578 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Ever tested for HIV | 9 months
  Binary endpoint: participant has ever tested for HIV vs. has never tested for HIV
Recent HIV testing | 9 months
  Binary endpoint: participant has tested since enrollment in the HIV trial vs. participant has not tested since enrollment in the HIV trial

SECONDARY OUTCOMES:
Use of HIV self-test | 9 months
  Binary outcome: participant has used HIV self-test since enrollment in the HIV trial vs. participant has not used an HIV self-test since enrollment in the HIV trial
Repeated HIV testing | 9 months
  Binary outcome: having tested at least twice since enrollment in the HIV trial vs. having tested once or fewer times since enrollment in the HIV trial
HIV status knowledge | 9 months
  Binary outcome: participant reports that he/she knows his/her HIV status
Correct report of HIV status | 9 months
  Binary outcome: participant correctly reports HIV status evaluated against biomarker HIV status vs. participant does not know or correctly report HIV status
Use of home rapid HIV test | 9 months
  Binary outcome: participant has used a rapid HIV test at home since enrollment in the HIV trial vs. particpant has not used rapid HIV test since enrollment in the HIV trial
HIV testing at healthcare facility | 9 months
  Binary outcome: participant has tested for HIV at a facility since enrollment in the HIV trial vs. participant has not tested for HIV at a facility since enrollment in the HIV trial
Linkage to HIV treatment and care | 9 months
  Binary outcome: participant has ever visited a facility where HIV treatment and care is available vs. participant has never visited a facility where HIV treatment and care is available
Recent linkage to HIV treatment and care | 9 months
  Binary outcome: participant has visited a facility where HIV treatment and care is available since enrollment in the HIV trial vs. participant has not visited a facility where HIV treatment and care is available since enrollment in the HIV trial
Number of recent sex partners | 9 months
  Count variable: number of sex partners since enrollment in the HIV trial
Recent condom use | 9 months
  Binary variable: participant has used condom with most recent sex partner vs. participant has not used condom with most recent sex partner
Most recent sex partner was casual or anonymous | 9 months
  Binary variable: most recent sex partner was casual or anonymous vs. most recent sex partner was neither casual nor anonymous
Rapid HIV testing during HAALSI | 9 months
  Binary outcome: participant used a rapid HIV test as part of the field operations of the mother study (HAALSI) since enrollment in the HIV trial vs. participant did not use an HIV test as part of the mother study since enrollment in the HIV trial
HIV treatment uptake | 9 months
  Binary outcome: participant has started HIV treatment vs. participant has not started HIV treatment
Antihypertensive treatment | 9 months
  Binary outcome: participant is currently receiving antihypertensive treatment vs. participant is currently not receiving antihypertensive treatment
Diabetes treatment | 9 months
  Binary outcome: participant currently receives diabetes treatment vs. participant currently does not receive diabetes treatment
Satisfaction with the fieldworker visit | 9 months
  Scale
Satisfaction with the South African government and healthcare system | 9 months
  Scale
Trust in other people and healthcare providers | 9 months
  Scale
Depressive Symptoms | 9 months
  CESD Scale
Viral load | 18-24 months
  Continuous variable: viral load
Blood pressure | 18-24 months
  Continuous outcome: blood pressure, systolic and diastolic
Blood sugar | 18-24 months
  Continous outcome: glucose or hemoglobin A1c
Biological Antiretroviral Screening | 18-24 months
  Binary Outcome: Presence of ART in blood

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, MD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- MRC/Wits Rural, Public Health and Health Transitions Research Unit (Agincourt), Acornhoek, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measures will be made available. Investigators from institutions outside those listed in this registration will be requested to obtain ethics permissions or exemptions for any analyses using these data from their institutional review boards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by the publication committee of the mother study (HAALSI). Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Gomez-Olive FX, Montana L, Wagner RG, Kabudula CW, Rohr JK, Kahn K, Barnighausen T, Collinson M, Canning D, Gaziano T, Salomon JA, Payne CF, Wade A, Tollman SM, Berkman L. Cohort Profile: Health and Ageing in Africa: A Longitudinal Study of an INDEPTH Community in South Africa (HAALSI). Int J Epidemiol. 2018 Jun 1;47(3):689-690j. doi: 10.1093/ije/dyx247. No abstract available. PMID 29325152